CLINICAL TRIAL: NCT02319174
Title: Accuracy Assessment of an Automatic Blood Pressure Measurement Device in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Marsh Rice University (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Rebecca Richards-Kortum, Stanley C. Moore Professor of Bioengineering, William Marsh Rice University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 14-082F-B
Record Dates: First submitted 2014-12-10; First posted 2014-12-18 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Pre Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sphygmo (Experimental): All subjects will have blood pressure measured by both the research device (Sphygmo) and the commercially available device. All clinical decisions will be made using measurements from the commercially available device.
  Interventions: Device: Sphygmo

INTERVENTIONS:
Device: Sphygmo — A team of engineers from Rice University has recently developed Sphygmo, an ambulatory, low-cost blood pressure monitor for use in the diagnosis and management of pre-eclampsia in low-resource hospitals

SUMMARY:
The purpose of the study is to help make a lower cost automatic blood pressure monitor device for diagnosis and monitoring of pre-eclampsia in pregnant women, where automatic blood pressure monitoring is limited or not available. The study will compare this low cost device to a commercially available system used for pre-eclamptic women in many United States hospitals that the investigators will be bringing to Malawi as a part of this study.

The team hopes to show that this lower cost blood pressure machine works well and can help women with pre-eclampsia. The study also aims to see if this machine is easy for the nurse to use.

70 pregnant women who are either at-risk or diagnosed with pre-eclampsia will be enrolled at University of Texas Health Science Center Houston. Patient arm circumference will be measured with measurement tape.

They will be seated upright in a comfortable chair with arm at heart level and an arm blood pressure cuff from either the automatic blood pressure monitor or a manual sphygmomanometer will be placed on the left arm.

The cuff will be inflated and then deflated until measurement concludes. Heart rate will be measured with tactile arterial palpation.The process will be repeated for a total of up to nine measurements, alternating between measurements with the automatic blood pressure monitor and the manual sphygmomanometer. There will be a waiting period of 45-60 seconds between each measurement.

The results of this study will help researchers understand the performance and usability of this device in Malawi and help decide if any design changes are needed.

DETAILED DESCRIPTION:
The research team has developed an automatic blood pressure monitor to be used for the monitoring and diagnosis of pre-eclampsia in pregnant women, particularly in low-resource settings where current monitoring is limited. This study aims to evaluate the accuracy of the device's blood pressure measurements in pregnant and pre-eclamptic women. This device must be evaluated with the above described population because blood pressure measurement devices are known to perform differently in pregnant and pre-eclamptic women than in normal healthy adults.

This study will take place at the University of Texas Health Science Center (UTHSC) where up to 70 subjects will be recruited to participate during their regularly scheduled antenatal care checkups.

1. The Patient arm circumference will be measured with measurement tape.
2. The Patient will be seated upright in a comfortable chair with arm at heart level.
3. An arm blood pressure cuff from either the automatic blood pressure monitor or a manual sphygmomanometer will be placed on the left arm of the patient over the brachial artery.
4. Cuff will be inflated to ~200 mmHg and then deflated until measurement concludes.
5. Heart rate will be measured with Tactile Arterial Palpation.
6. Steps 3-4 will be repeated for a total of up to nine measurements, alternating between measurements with the automatic blood pressure monitor and the manual sphygmomanometer. There will be a waiting period of 45-60 seconds between each measurement.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women receiving antenatal care at the UT OB/GYN clinic.
* Over the age of 18

Exclusion Criteria:

* Women under the age of 18
* Women unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca R Kortum, PhD, Principal Investigator — William Marsh Rice University
Locations (1):
- University of Texas Health Science Center Houston, Houston, Texas, United States

REFERENCES:
- [Background] Natarajan P, Shennan AH, Penny J, Halligan AW, de Swiet M, Anthony J. Comparison of auscultatory and oscillometric automated blood pressure monitors in the setting of preeclampsia. Am J Obstet Gynecol. 1999 Nov;181(5 Pt 1):1203-10. doi: 10.1016/s0002-9378(99)70109-2. PMID 10561646
- [Background] Turner JA. Diagnosis and management of pre-eclampsia: an update. Int J Womens Health. 2010 Sep 30;2:327-37. doi: 10.2147/IJWH.S8550. PMID 21151680
- [Background] Dekker G, Sibai B. Primary, secondary, and tertiary prevention of pre-eclampsia. Lancet. 2001 Jan 20;357(9251):209-15. doi: 10.1016/S0140-6736(00)03599-6. PMID 11213110
- [Background] Magee LA, Abalos E, von Dadelszen P, Sibai B, Easterling T, Walkinshaw S; CHIPS Study Group. How to manage hypertension in pregnancy effectively. Br J Clin Pharmacol. 2011 Sep;72(3):394-401. doi: 10.1111/j.1365-2125.2011.04002.x. PMID 21545480
- [Background] De Greeff A, Ghosh D, Anthony J, Shennan A. Accuracy assessment of the Dinamap ProCare 400 in pregnancy and preeclampsia. Hypertens Pregnancy. 2010 Jan;29(2):198-205. doi: 10.3109/10641950902968650. PMID 20367507
- [Background] O'Brien E, Petrie J, Littler W, de Swiet M, Padfield PL, Altman DG, Bland M, Coats A, Atkins N. An outline of the revised British Hypertension Society protocol for the evaluation of blood pressure measuring devices. J Hypertens. 1993 Jun;11(6):677-9. doi: 10.1097/00004872-199306000-00013. No abstract available. PMID 8397248

RESULTS

PARTICIPANT FLOW:
Groups:
- Sphygmo: All subjects will have blood pressure measured by both the research device (Sphygmo) and the commercially available device. All clinical decisions will be made using measurements from the commercially available device. All subjects are pregnant women.
  Sphygmo: A team of engineers from Rice University recently developed Sphygmo, an ambulatory, low-cost blood pressure monitor for use in the diagnosis and management of pre-eclampsia in low-resource hospitals
Period: Overall Study
Arm/Group | Sphygmo
Started | 43
Completed | 42
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Sphygmo: All subjects will have blood pressure measured by both the research device (Sphygmo) and the commercially available device. All clinical decisions will be made using measurements from the commercially available device. All subjects are pregnant women.
  Sphygmo: A team of engineers from Rice University has recently developed Sphygmo, an ambulatory, low-cost blood pressure monitor for use in the diagnosis and management of pre-eclampsia in low-resource hospitals
Arm/Group | Sphygmo
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 29 [18 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Blood Pressure Readings by Sphygmo
Description: Mean difference of systolic and diastolic blood pressures between Sphygmo blood pressure measurements and measurements from the gold standard sphygmomanometer.
Time Frame: Blood pressure was measured an average of 9 times for each participant and the average of these measurements was recorded. Each measurement period lasted approximately 30-45 minutes
Population: Of 41 participants who completed the study, 5 participants were excluded on account of the observer reporting a difficulty in hearing, movement, or uncertainty with the measurement. This left 36 participants, 18 of which were used to train the device. The data presented here is from the remaining 18 participants.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Dinamap: All subjects will have blood pressure measured by both the research device (Sphygmo) and the commercially available device. All clinical decisions will be made using measurements from the commercially available device. All subjects are pregnant women.
  Dinamap: Dinamap is a commercially available, ambulatory, blood pressure monitor for use in the diagnosis and management of pre-eclampsia in low-resource hospitals
Arm/Group | Sphygmo | Dinamap
Number analyzed (Participants) | 18 | 18
mmHg
  Systolic Mean | 114.5 (10.9) | 115.6 (12.5)
  Diastolic Mean | 65.7 (8.3) | 66.3 (10.6)

2. Primary Outcome: Percent of Sphygmo Readings That Were Within 5mmHg, 10mmHg, and 15mmHg of the Readings by the Gold Standard Sphygmomanometer.
Description: The British Hypertension society defines a specific criteria for the accuracy of a sphygmomanometer. Devices are graded according to the cumulative percentage of readings that have an absolute difference between the more favorable observer's mercury sphygmomanometer readings and the test device of < 5 mmHg, < 10 mmHg, and < 15 mmHg. A letter grade of "A" requires that over 60%, 85%, and 95% were achieved in the < 5 mmHg, < 10 mmHg, and <15 mmHg categories, respectively. A letter grade of "B" requires that over 50%, 75%, and 90% were achieved in the < 5 mmHg, < 10 mmHg, and <15 mmHg categories, respectively. The test device achieved a grade of (A/A) with the validation data from this study.
Time Frame: Blood pressure was measured an average of 9 times for each participant during their single measurement period, and the average of those measurements was recorded. Each measurement period lasted approximately 30-45 minutes
Population: as for outcome 1
Measure: Number; unit: percentage of measurements in range
Arm/Group | Sphygmo
Number analyzed (Participants) | 18
percentage of measurements in range
  Systolic Difference <5 mmHg | 67
  Systolic Difference <10 mmHg | 85
  Systolic Difference <15 mmHg | 98
  Diastolic Difference <5 mmHg | 70
  Diastolic Difference <10 mmHg | 89
  Diastolic Difference <15 mmHg | 98

ADVERSE EVENTS:
Time Frame: 1 year and 5 months.
Arm/Group | Sphygmo
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No